CLINICAL TRIAL: NCT01463943
Title: "An Open-Label, Non-Inferiority, Phase III Trial Comparing Eurofarma's Experimental Product Saccharomyces Boulardii Versus Floratil® (S. Boulardii - Merck) in the Prevention of Antibiotic-Associated Diarrhea."
Brief Title: Non-Inferiority Trial Comparing Eurofarma's Experimental Product Saccharomyces Boulardii Versus Floratil® in the Prevention of Antibiotic-Associated Diarrhea
Acronym: ACROSS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change company strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EF 121
Record Dates: First submitted 2011-10-27; First posted 2011-11-02 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2011-10

CONDITIONS: Antibiotics
MeSH Terms: interventions — Probiotics

ARMS (3):
- Saccharomyces boulardii capsules (200 mg). (Experimental)
  Interventions: Other: Probiotic
- Floratil® (Active Comparator)
  Interventions: Other: Probiotic
- Saccharomyces boulardii powder (200 mg). (Experimental)
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Probiotic
  Arms: Saccharomyces boulardii capsules (200 mg).
Other: Probiotic
  Arms: Saccharomyces boulardii powder (200 mg).
Other: Probiotic
  Arms: Floratil®

SUMMARY:
The study's objective is to evaluate the efficacy and safety of two formulations for the prophylactic treatment of diarrhea in subjects using antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. ICF signature;
2. The subject must agree to follow the instructions and to perform study procedures and visits;
3. Male and female subjects between 18 and 65 years old;
4. Subjects who have scheduled a treatment or started the use of antibiotics over 24 hours ago:

Exclusion Criteria:

1. Generalized infection or bacteremia;
2. Chronic gastrointestinal diseases (e.g., Crohn's Disease and Irritable Bowel Syndrome);
3. Documented chronic diarrhea;
4. Acute diarrhea episode within 24 hours prior to the start of antibiotic use. Use of tube feeding (nasogastric and nasoenteral);
5. Immunodeficiency (radiotherapy or chemotherapy);
6. Use of food with probiotic properties in the last 10 days;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
frequency of diarrhea in subjects using antibiotics

SECONDARY OUTCOMES:
Frequency of diarrhea by severity

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernando Francesconi, MD, Principal Investigator — Hospital Mãe de Deus; Flavio Quillici, MD, Principal Investigator — UNIGASTRO; Martti Antila, MD, Principal Investigator — Clínica de Alergia Martti Antila; Olavo Mion, MD, Principal Investigator — Hospital das Clínicas - SP; José Angelo Rizzo, MD, Principal Investigator — Universidade Federal de Pernambuco; Carlos Cezar Fritscher, MD, Principal Investigator — Hospital São Lucas da PUC - RS; Ronaldo Damião, MD, Principal Investigator — Hospital Universitario Pedro Ernesto; Flávio Steinwurtz, MD, Principal Investigator — Hospital Albert Einstein; Cyrla Zaltman, MD, Principal Investigator — Hospital Universitário Clementino Fraga Filho; José Hungria Neto, MD, Principal Investigator — Santa Casa de Misericórdia; Newton Carvalho, MD, Principal Investigator — Hospital de Clínicas da Universidade Federal do Paraná; Julio Cesar Teixeira, MD, Principal Investigator — University of Campinas, Brazil; Andreia Luisa Francisco Pez, MD, Principal Investigator — Pesquisare Saúde S/S Ltda; Paola Colares de Borba, MD, Principal Investigator — Instituto de Prevenção ao Câncer do Ceará; Cecília Roteli Martins, MD, Principal Investigator — HOSPITAL MATERNIDADE LEONOR MENDES DE BARROS; Paulo Sérgio Viero Naud, MD, Principal Investigator — Hospital das Clínicas de Porto Alegre; Bruno Gonçalves, MD, Principal Investigator — Hospital Leforte
Locations (17):
- Brazil (17):
  - UNICAMP, Campinas
  - Unigastro, Campinas
  - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba
  - Instituto de Prevenção ao Câncer do Ceará, Fortaleza
  - Hospital das Clinicas de Porto Alegre, Por to Alegre
  - Hospital São Lucas da PUC - RS, Porto Alegre
  - Mãe de Deus Center, Porto Alegre
  - Universidade Federal de Pernambuco, Recife
  - Hospital Universitário Clementino Fraga Filho (UFRJ), Rio de Janeiro
  - Hospital Universitário Pedro Ernesto, Rio de Janeiro
  - Pesquisare Saúde S/S Ltda, Santo André
  - Hospital Albert Einstein, São Paulo
  - Hospital das Clínicas, São Paulo
  - Hospital Leforte, São Paulo
  - Hospital Maternidade Leonor Mendes de Barros, São Paulo
  - Santa Casa de Misericórdia, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba